CLINICAL TRIAL: NCT06284304
Title: A Pilot Study of Dose dE-eScalaTion IN prostATe radIOtherapy usiNg the MRL
Acronym: DESTINATION
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N22DES
Record Dates: First submitted 2024-02-05; First posted 2024-02-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer
Keywords: Radiotherapy; De-escalation; Prostate cancer; MR-Linac
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental radiotherapy treatment (Experimental): SBRT 5x30Gy of whole prostate and isotoxic 45 Gy GTV plus intra-prostatic margin
  Interventions: Radiation: De-escalated radiotherapy

INTERVENTIONS:
Radiation: De-escalated radiotherapy — 5 fraction de-escalated dose SBRT protocol

SUMMARY:
Trial design: A single centre phase II non-randomised study

Trial population: Men with intermediate risk localised prostate cancer

Recruitment target: 20 patients in total

Trial objectives:

* Primary To develop a 5 fraction de-escalated dose SBRT protocol capable of reducing side effects
* Secondary

  * To assess levels of acute GU and GI toxicity (CTCAE)
  * To assess levels of late GU and GI toxicity (CTCAE)
  * To assess late sexual quality of life (expanded EPIC, IIEF-5)
  * To assess biochemical relapse-free survival at 2 years

Trial treatment: All radiotherapy will be delivered on the MR-linac. Intraprostatic dose will be varied according to risk of local recurrence, based on mpMRI, PSA and histology. The whole prostate will receive 30 Gy in 5 fractions and the GTV plus intra-prostatic margin will receive an isotoxic 45 Gy prescription.

DETAILED DESCRIPTION:
Primary endpoint: Technical feasibility of treating prostate cancer with toxicity- minimising radiotherapy on an MR-linac

Secondary endpoint:

* Physician reported GU and gastrointestinal (GI) toxicity (CTCAE grade) at baseline and the end of treatment then at 4 weeks and 3 months post-treatment.
* Late toxicity (CTCAE v5.0) at 1 and 2 years post-treatment
* Patient-reported outcome measures (PROMs) from the EPIC-26, IPSS, and IIEF-5 questionnaires. Patients will be asked to complete PROMs at 4 weeks, 3 and 6 months, 1 and 2 years post treatment.
* PSA control and kinetics at 2 years post-treatment

Quality of life: EPIC-26 QoL will be measured at baseline, then at 4 weeks and 3, 6, 12 and 24 months from end of treatment. IIEF-5 will be completed at baseline and months 6, 12 and 24. IPSS will be measured at all time points.

Follow-up: Patients will be assessed at 6, 12 and 24 months and then as per standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged ≥18 years
2. Histological confirmation of prostate adenocarcinoma requiring radical radiotherapy
3. Gleason score 3+3, 3+4 or 4+3 (Grade groups 1, 2 or 3)
4. MRI stage T2 or less (as staged by AJCC TNM 2018)
5. MRI-visible tumour(s) of PIRADS v2 grade 3 or higher on T2 and diffusion-weighted imaging and/or dynamic contrast-enhanced imaging with concordant pathology
6. Dominant lesion <50% of prostate on any axial slice and <50% total prostate volume
7. PSA <20 ng/ml prior to starting ADT
8. Patients can be concurrently treated with androgen deprivation therapy if this would be standard of care. LHRH analogues or Bicalutamide are permitted. ADT is not mandatory where this would usually be omitted.
9. WHO Performance status 0-2
10. Ability of the participant understand and the willingness to sign a written informed consent form.
11. Ability/willingness to comply with the patient reported outcome questionnaires schedule throughout the study.

Exclusion Criteria:

1. Contraindications to MRI (e.g. pacemaker, potentially mobile metal implant, claustrophobia)
2. IPSS 19 or higher
3. High grade disease (GG3) occult to MRI-defined lesion
4. Post-void residual >100 mls, where known
5. Prostate volume >90cc
6. Comorbidities which predispose to significant toxicity (e.g. inflammatory bowel disease) or preclude long term follow up
7. Unilateral or bilateral total hip replacement, or other pelvic metalwork which causes artefact on diffusion-weighted imaging
8. Previous pelvic radiotherapy
9. Patients needing >6 months of ADT due to disease parameters.
10. Previous invasive malignancy within the last 2 years excluding basal or squamous cell carcinomas of the skin, low risk non-muscle invasive bladder cancer (assuming cystoscopic follow up now negative) or small renal masses on surveillance

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04-02 (Estimated)

PRIMARY OUTCOMES:
Technical feasibility of treating prostate cancer with toxicity minimising radiotherapy on a MR-linac | after 1,5 week of treatment
  To establish the technical feasibility of treating prostate cancer with tumour-escalated/normal prostate de-escalated dose radiotherapy on an MR-linac. Feasiblity is defined as coverage of GTV boost D90% >42Gy on the post-treatment imaging.

SECONDARY OUTCOMES:
Acute GU toxicity | within 90 days after first radiation treatment
  Physician-reported acute GU and GI toxicity according to the CTCAE v5.0.
Acute GI toxicity | within 90 days after first radiation treatment
  Physician-reported acute GU and GI toxicity according to the CTCAE v5.0.
Late GU toxicity | After at least 90 days after the first radioation treatment up to 2 years
  Physician-reported late GU and GI toxicity according to the CTCAE v5.0.
Late GI toxicity | After at least 90 days after the first radioation treatment up to 2 years
  Physician-reported late GU and GI toxicity according to the CTCAE v5.0.
PROMs | 2 years
  will be assessed using the International Prostate Symptom Score (IPSS) questionnaire, the EPIC-26 questionnaire and the IIEF-5 questionnaire.
Biochemical free survival | Up to 2 years
  PSA control, biochemical failure/progression. Biochemical failure is defined a PSA nadir+ 2 ng/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Floris Pos, MD PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No